CLINICAL TRIAL: NCT07383727
Title: Readiness to Change and the Implementation of Home Modifications for Adults Over 60
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University of Vermont (Other)
Responsible Party: Principal Investigator, Victoria Priganc, Associate Professor, University of Vermont
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Other
Other Study IDs: IRB00003816
Record Dates: First submitted 2026-01-26; First posted 2026-02-03 (Actual); Last update posted 2026-02-03 (Actual); Status verified 2026-01

CONDITIONS: Older Adults (60 - 85 Years Old)
Keywords: readiness to change; home modifications; older adults; aging-in-place

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- face-to-face education (Other): This group will receive face-to-face education regarding home modifications.
  Interventions: Other: Face-to-face educational session
- on-line education (Other): This group will receive on-line education regarding home modifications.
  Interventions: Other: On-line educational session

INTERVENTIONS:
Other: Face-to-face educational session — Subjects will receive face-to-face education regarding different home modifications.
  Arms: face-to-face education
Other: On-line educational session — Subjects will watch an on-line video describing different home modifications.
  Arms: on-line education

SUMMARY:
This study is focused on home modifications and the changes that older adults may experience while aging. We are conducting this study to better understand how people feel about making changes to their homes or utilizing equipment to assist with home tasks.

DETAILED DESCRIPTION:
Understanding people's readiness for change could be used as a predictor of an older adult's willingness to implement home modifications to improve aging in place and safety. Adults benefit from home modifications as they age but are often hesitant to make these changes despite support from occupational therapists and other healthcare initiatives. Some benefits of home modifications include reduced fall risk and depression, and increased independence in activities of daily living. The readiness to change scale has been used in multiple areas of older adult research to understand health behavior change including physical activity, driving cessation, and functional activities. We are therefore investigating what relationship lies between readiness to change scale, methods of delivering education around the importance of home modifications, and adoption of home modifications in older adults.

Subjects 60 or older who are living independently will be recruited through the investigator's network of clinical providers, the Vermont Older Adult Research Registry, and through various community organizations that address the needs of older adults.

Subjects will be contacted via phone or in-person. Inclusion/exclusion criteria will be discussed with those expressing an interest in the study. Subjects that meet the inclusion exclusion criteria will be invited to participate in the study.

* Obtaining consent for subjects via phone recruitment: For those subjects who express an interest via a phone call, a RedCap link will be sent via email. The RedCap link will have the consent form and at the end, a place for an electronic signature. This phone call and review of consent form will be conducted by the research team.
* Obtaining consent for subjects via in-person: For those subjects who express an interest via an in-person meeting, a member of the research team will review the consent form and a consent signature will be gathered after review of the study.

Once subjects consent to participate in the study, subjects will be randomly assigned using a random number generator to the face-to-face group or the online group.

Face-to-face group: Once assigned, subjects will be invited to the face-to-face session via three avenues. 1) the research team can meet the individual in their home, 2) the subject can come to the UVM Occupational Therapy Smart Apartment lab, 3) the subject can come to a community center. Sessions in the UVM Occupational Therapy Smart Apartment lab and the community centers may be group sessions or individual sessions. To start the session, subjects will complete a demographic intake form, the readiness to change scale, and a home modification survey. These surveys will be paper surveys. Next, the research team will offer a hands-on educational session describing the benefits of home modifications and allowing participants to trial different devices. Following the hands-on education session, subjects will be asked to again complete the readiness to change scale and the home modification survey. The entire time commitment will be approximately 1-hour.

Online group: Once assigned, subjects will be sent a Qualtrics link that contains the demographic intake form, the readiness to change scale, and home modification survey. These surveys will be done on-line via Qualtrics. Subjects will be asked to complete the initial paperwork within 7 business days of consenting to participate in the study. The research team will reach out to the participants after 7 days to ensure the initial paperwork has been completed. Once the intake form and surveys have been completed, a zoom meeting will be set up to explain how they can view the educational session and to talk about some challenges they have in their homes. Subjects will then be given a link to an educational session on a private YouTube channel. They can watch the educational session at a time of their convenience, but will be asked to complete it within 10-14 business days from completing the initial intake form and surveys. The educational video should take no longer than 30-minutes to watch. Once completed, they will be encouraged to reach out to the research team with questions. The researchers will reach out at 10-14 business days to see if there are any questions or if they have completed the on-line educational session. At that point, participants will be sent another Qualtrics link to complete the post-surveys (readiness to change scale and home modification survey).

All subjects regardless of group assignment will be followed-up via a phone call 3-months later to identify if any modifications have been implemented. The same phone script will be used and all data gathered from the 3-month follow-up will be gathered via a phone call.

ELIGIBILITY:
Inclusion Criteria:

* Adults over 60
* Living independently
* Able to read, speak, understand English

Exclusion Criteria:

* Individuals unable to legal represent themselves

Min Age: 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Estimated)
Dates: Start 2026-01-28 (Estimated); Primary Completion 2026-06-30 (Estimated); Study Completion 2026-06-30 (Estimated)

PRIMARY OUTCOMES:
Readiness to change scale | From enrollment to the end of treatment at 1 day - 10 days.

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Dermody G, Fritz R, Glass C, Dunham M, Whitehead L. Factors influencing community-dwelling older adults' readiness to adopt smart home technology: A qualitative exploratory study. J Adv Nurs. 2021 Dec;77(12):4847-4861. doi: 10.1111/jan.14996. Epub 2021 Sep 3. PMID 34477222
- [Background] Mark JA, Henry A, Moreland B, Dobash D, Bergen G. Assessing Older Adults' Readiness for Adopting Fall Prevention Recommendations Using the Transtheoretical Stages of Change. J Appl Gerontol. 2025 May;44(5):726-736. doi: 10.1177/07334648241289933. Epub 2024 Oct 22. PMID 39439095
- [Background] Rose KC, Gitlin LN, Dennis MP. Readiness to use compensatory strategies among older adults with functional difficulties. Int Psychogeriatr. 2010 Dec;22(8):1225-39. doi: 10.1017/S1041610210001584. Epub 2010 Jul 27. PMID 20663239